CLINICAL TRIAL: NCT02967900
Title: Longitudinal Study of Chronic Wounds Using Novel Wound Measurement Technologies
Status: Completed | Type: Observational
Sponsor: Michelson Diagnostics Ltd. (Industry)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1200
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — 2 mm punch biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An open, non-randomised longitudinal study of diabetic foot ulcers receiving standardised treatment, over a 16 week period conducted at out-patient level, utilising novel optical wound measurement technologies.

DETAILED DESCRIPTION:
Diabetic foot ulcers are a major burden on the healthcare system, and it is highly desirable to develop a practical, reliable, non-invasive means of diagnosing, assessing and measuring wound healing, so as to provide wound care specialists with key data with which to make effective decisions for clinical management.

Optical coherence tomography (OCT) is a novel technique of imaging of cutaneous tissue. Using low-power infrared light, it is a non-invasive in-vivo imaging technique which provides resolution of <10microns to a depth of 1 - 1.25 mm in skin, (adequate to resolve capillaries) utilizing the optical scattering characteristics of tissue to provide imaging contrast.

This open, non-randomised, observational study will assess the feasibility of using OCT to diagnose chronic diabetic foot ulcers. One cohort of 15 patients will be scanned over a 16 week period and results studied to determine whether there is an association between rate of wound healing and OCT measurements.

ELIGIBILITY:
Inclusion Criteria:

* Defining ABPI ≥0.5 - <1.2
* Patients with DFU for over 4 weeks but less than 1 year duration. DFU resulting from neuropathy will be included.
* Neuropathy scores defined by 10g Semmes-Weinstein monofilament tests at 10 sites on plantar and dorsal surfaces

Exclusion Criteria:

* Patients with uncontrolled diabetes, the Charcot Foot, cancer (except non-melanoma skin cancer in the limb), decompensated cardiac failure, clinically significant renal failure, history of stroke or significant peripheral arterial disease, or those who are pregnant, or on a waiting list for interventional therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending hospital outpatient, day care or inpatient clinic, > 18 years and capable of giving informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Correlation of OCT Measurement of blood vessel density with rate of wound healing | 16 weeks
  Pearson's coefficient of correlation between the OCT measurement of blood vessel density (fraction of the imaged skin volume in the upper 0.5 mm of tissue that is comprised of vessels with detectable blood flow) and the rate of wound healing (defined as the magnitude of reduction in measured area of the wound per 4 week period), as an average across all trial subjects and all measurement points during the trial.
  Pearson's coefficient > 50% signifies a positive result.

SECONDARY OUTCOMES:
Correlation of OCT Measurement of blood vessel density at baseline, with rate of wound healing | 16 weeks
  Pearson's coefficient of correlation between the OCT measurement of blood vessel density at baseline, (fraction of the imaged skin volume in the upper 0.5 mm of tissue that is comprised of vessels with detectable blood flow), and the rate of wound healing (defined as the magnitude of reduction in measured area of the wound over the 16 week trial period), as an average across all trial subjects.
  Pearson's coefficient > 50% signifies a positive result.

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Bowling, PhD, Principal Investigator — Central Manchester University Hospital NHS Foundation Trust
Locations (1):
- Manchester Royal Infirmary, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No